CLINICAL TRIAL: NCT04065334
Title: Effects of Low- Versus High Dose High Intensity Interval Training and Strength Training on Physical Health in Substance Use Disorder Patients: A Randomized Controlled Trial
Brief Title: Exercise Training as Medicine for Substance Use Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/502
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders
Keywords: Resistance training; Endurance training
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose training (Experimental)
  Interventions: Behavioral: low dose training
- high dose training (Active Comparator)
  Interventions: Behavioral: High dose training

INTERVENTIONS:
Behavioral: High dose training — 4 x 4 minutes of high intensity workload on treadmill and 4 repetitions x 4 sets of high intensity workload in hack squat
  Arms: high dose training
Behavioral: low dose training — 1 x 4 minutes of high intensity workload on treadmill and 2 repetitions x 4 sets of high intensity workload in hack squat
  Arms: low dose training

SUMMARY:
This study compares the effects of high dose and low dose, high intensity, endurance training and strength training in substance use disorder patients. The hypothesis is that the increase in endurance (measured as maximal oxygen uptake) and strength (measured as maximal strength) will be similar in both the high dose and low dose training groups after 24 training sessions over eight weeks. The rationale for this assumption is based on the patient groups poor physical capacity, supporting that a lesser physical workload is needed to achieve a substantial increase in physical capacity. The practical implication could be higher training attendance, because it is likely easier to motivate the patient group when they only have to perform half the workload. It is paramount for this patient group to increase their physical capacity and consequently augment their physical health status since they are in a high-risk group for developing life-threatening lifestyle related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being an inpatient at the clinic
* Free of known cardiovascular disease, pulmonary disease and cancer

Exclusion Criteria:

* Not able to perform a maximal treadmill test
* Not able to perform a maximal strength test in hack squat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
change in oxygen uptake | baseline to 8 weeks
  cardiopulmonary exercise test (CPET) objective gas measurements
change in leg muscular strength | baseline to 8 weeks
  One repetition maximum strength test half squat

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Smedsrud, Study Director — St. Olavs Hospital
Locations (1):
- Klinikk for rus- og avhengighetsmedisin, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loe H, Mosti MP, Wisloff U, Haberstroh C, Flemmen G. Cardiopulmonary and muscular effects of different doses of high-intensity physical training in substance use disorder patients: study protocol for a block allocated controlled endurance and strength training trial in an inpatient setting. BMJ Open. 2022 Sep 27;12(9):e061014. doi: 10.1136/bmjopen-2022-061014. PMID 36167363